CLINICAL TRIAL: NCT00635076
Title: A Randomized, Double-blind, Placebo-controlled Study of Continuation Treatment With Xanax XR in the Treatment of Adolescents With a Primary Diagnosis of Panic Disorder
Brief Title: A Study to Assess the Long-term Use of Alprazolam Extended Release (XL) in the Treatment of Adolescents With Panic Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Please see Detailed Description for the termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6131007
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Other: placebo
- Alprazolam XR group (Active Comparator)
  Interventions: Drug: alprazolam XR

INTERVENTIONS:
Other: placebo — Patients continued taking the matching placebo that they were taking when they completed Study A6131002 (oral tablets taken once daily).
  Arms: Placebo group
Drug: alprazolam XR — Patients continued taking the same dosage of alprazolam that they were taking when they completed Study A6131002 (oral tablets taken once daily (1-6mg)); patients taking less than 6 mg/day who failed to show a satisfactory clinical response since the previous visit, and who were free of dose-limiting adverse events, could have their dosage titrated upward by 1 mg/day; upward daily dosage titration of 1 mg was allowed every 7 days, up to a maximum daily dosage of 6 mg/day; patients who were unable to tolerate the previous dosage level of alprazolam XR could have their daily dosage reduced.
  Other Names: Xanax XR
  Arms: Alprazolam XR group

SUMMARY:
The purpose of this study is to evaluate the long-term (6-month) efficacy, safety, and tolerability of alprazolam XR in adolescents with panic disorder.

DETAILED DESCRIPTION:
Due to recruitment difficulties in this adolescent population, the clinical program for alprazolam XR was cancelled and this study was terminated on 1 September 2004. There were no safety concerns that led to this decision.

ELIGIBILITY:
Inclusion Criteria:

* A primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision diagnosis of panic disorder with or without agoraphobia based on the Mini-International Neuropsychiatric Interview for Children and Adolescents
* Subjects with an average of 1) at least one 4-symptom panic attack per week over the last 4 weeks before screening; 2) at least one 4-symptom panic attack per week over the last 4 weeks before baseline; and 3) at least one 4-symptom panic attack in the 7 days prior to baseline
* To enter Study A6131007, subjects must have completed Study A6131002, had an acceptable tolerability to study drug, and in the clinical judgment of the investigator, could have benefited from continued study treatment.

Exclusion Criteria:

* Subjects must continue to meet all of the exclusion criteria enumerated in the Acute Efficacy Study (Protocol A6131002) with the following exception: Subjects will be allowed to undergo cognitive-behavioral or other panic-specific therapy and any other psychotherapy (e.g., supportive and/or family therapy) during the expected study period in this study.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2004-07; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Baseline-to-peak Physician Withdrawal Checklist change score during taper off Alprazolam | Week 24 (taper baseline), Weeks 25-29, and end of taper visit
The incidence of treatment-emergent adverse events during 6 months of treatment with alprazolam XR | Weeks 6, 8, 12, 16, 20, and 24
Endpoint change from baseline in Digit Symbol-Coding Test, immediate recall, and delayed recall | Week 24

SECONDARY OUTCOMES:
Endpoint change from baseline in Hamilton Anxiety Rating scale | Weeks 12 and 24
Endpoint change compared with baseline in the Panic Disorder Severity Scale - Adolescent Version total and item scores | Weeks 12 an 24
Endpoint compared with baseline for Clinical Global Impression (CGI)-Improvement scale | Weeks 12 and 24
Endpoint change compared with baseline in CGI-Severity score | Weeks 12 and 24
Endpoint compared with baseline in Pediatric Quality of Life, Enjoyment, and Satisfaction Questionnaire improvement score | Weeks 12 and 24
Descriptive estimates of the persistence of safety events and adverse events | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Middleton, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131007&StudyName=A%20study%20to%20assess%20the%20long-term%20use%20of%20alprazolam%20extended%20release%20%28XL%29%20in%20the%20treatment%20of%20adolescents%20with%20panic%20disorder